CLINICAL TRIAL: NCT00023465
Title: Quantification of Pulmonary Neutrophil Activity in Cystic Fibrosis Using Radiolabeled Fluorodeoxyglucose and PET Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-MO1RR00036-0798
Record Dates: First submitted 2001-09-06; First posted 2001-09-10 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: FDG-PET
Procedure: spirometry
Procedure: bronchoscopy with BAL

SUMMARY:
It has been shown that neutrophils (a specific type of cell) are involved in inflammation in the lungs of CF patients. Neutrophil levels in CF patients have been measured by bronchoalveolar lavage (BAL), which samples cells in the fluid lining of the lungs. Other studies have measured neutrophil levels and inflammation in other parts of the body using PET scanning. This study aims to show that PET scanning can be used as a non-invasive marker of inflammation in the lungs of patients with CF, which would be a useful tool in treatment.

The primary goal of this study is to draw a connection between the level of inflammation shown in the PET scan and the number of neutrophils obtained from the BAL. This study will also look at how the PET images relate to inflammatory molecules in the lungs and to the FEV-1 obtained through spirometry.

DETAILED DESCRIPTION:
All patients involved in the study will have a PET scan performed. This involves injecting a small amount of radiolabelled glucose (sugar) into the blood. A scan will then be performed to obtain an image of where in the body that glucose is being used. Patients will also have spirometry done. Spirometry is a simple procedure measuring the functioning of the lungs (FEV-1) by measuring the amount of air a patient can blow out and inhale (the patient breathes into a machine). Bronchoalveolar lavage (BAL) will be performed. This involves putting a small amount of fluid into a section of the lung, then suctioning it out to retrieve the cells and molecules contained in the substance lining the lung.

Subjects will be patients with cystic fibrosis. Ten subjects will be stable with either mild or moderate disease. These subjects will receive a PET scan, spirometry, and BAL.

This portion of the study is made up of 10 stable CF patients, 5 of whom will have mild disease, and 5 of whom will have moderate disease. These patients will receive a PET scan, spirometry and a BAL over 2 consecutive days. On day 1, patients will have a PET scan and spirometry. On day 2, patients will have a BAL.

Patients will arrive on the first day after fasting for at least 6 hours and will be taken to the PET facility. PET scanning consists of a 2-minute scan followed by a 15-minute scan, injection of radiolabelled sugar into the vein, and 66 minutes of scanning. The patient will then be instructed to empty his or her bladder to reduce total radiation exposure. The patient will then be given a meal. Next, the patient will be taken for spirometry, the last test of day 1, which simple involves breathing into a machine that measures the amount of air inhaled and exhaled. Upon reporting to the GCRC on day 2, the patient will be taken for a BAL (the patient will have fasted for at least 6 hours prior to admission). BAL involves a small tube placed into the mouth, down the throat, and into the lung (lidocaine is used to numb the entire area). Less than 3 tablespoons of saline (salt water) is poured down the tube, then immediately sucked back up and collected by the doctor. This is repeated twice, for a total of 8 tablespoons of liquid.

ELIGIBILITY:
Inclusion criteria:

1. Subject has Cystic Fibrosis
2. Subject must be capable of lying still and supine within the PET scanner for approximately 90 minutes.
3. Subject must be capable of fasting for 6 hours
4. Subjects must fall into one of the following three categories: Study 1 Group A: Stable Patient with mild CF. Must have an FEV1 of greater than 65% predicted. Study 1 Group B: Stable Patient with moderate/moderately severe CF. Must have an FEV1 of between 40% and 65% predicted. Study 2: Acutely Ill Patient: CF patient admitted to the hospital with acute exacerbation of obstructive lung disease associated with CF, requiring hospitalization.
5. Subjects in study 2 must be willing to return within 4 weeks for re-evaluation upon convalescence.
6. The treating physician has granted verbal permission for patient to participate in this study.
7. Subjects in study 2 will have had spirometry upon admission.

Exclusion Criteria:

1. Failure to obtain informed consent.
2. Pregnancy (confirmed by a qualitative urine hCG pregnancy test)
3. Lactation
4. Subject is enrolled in another study involving the use of radioisotopes or another research study of an investigational drug
5. For subjects in groups 1A and 1B, inability to tolerate BAL (ie, medically unstable)
6. Diagnosis of diabetes or fasting blood sugar >150 mg/dl
7. Study 1: FEV1 <40% predicted
8. Study 2: baseline (prehospitalization) FEV1 <40% predicted
9. Patient requires mechanical ventilation
10. Patient has received G-CSF (granulocyte colony stimulating factor) within the last 5 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States